CLINICAL TRIAL: NCT02830022
Title: Sleep, Autonomic Nervous System and Cardiorespiratory Capacity in Autism Spectrum Disorders Children
Brief Title: Sleep, Autonomic Nervous System and Cardiorespiratory Capacity in Autism Spectrum Disorders Children (APAUTRES)
Acronym: APAUTRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC14.123
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Autonomic Nervous System Diseases; Sleep
Keywords: autism spectrum disorder
MeSH Terms: conditions — Autonomic Nervous System Diseases; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Experimental): Children from 8 to 18 years with autism without without intellectual disabilities (IQ > 70), verbals and responding to classification CIM 10-DSM IV.
  Interventions: Other: physiological explorations
- Healthy volunteers (Experimental): Paired for age, gender, IQ and and the practice of a physical activity strictly within the school context.
  Interventions: Other: physiological explorations

INTERVENTIONS:
Other: physiological explorations

SUMMARY:
Autism Spectrum Disorders (ASD) is a neurodevelopmental disorder which involves social and behavioural impairments. Autonomic dysfunctions and disturbed sleep were often associated to ASD. The investigators proposed to explore the impact of physical activity on these disorders. In this context, it is necessary to characterize the cardiorespiratory capacities of ASD children in order to promote physical activity for this population. To examine potential differences between ASD and control children, some explorations were proposed: a maximal treadmill test, motor evaluation, and orthostatic test (for the evaluation of autonomic nervous system).

An actimetry during one week (evaluation of physical activity and sleep) completed this study in order to specify sleep characteristic and established the possible link between physical activity sleep characteristics and physical fitness in ASD children.

ELIGIBILITY:
Inclusion Criteria:

* children physically active
* children with an intellectual quotient >70
* for autism children a diagnosis of autism in accordance to DSMV

Exclusion Criteria:

* history of cardio-vascular disease
* history of asthma or respiratory disease
* Behavior disorders.
* medical treatment by neuroleptic or melatonin or antiepileptic

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2013-12-11 (Actual); Primary Completion 2017-06-11 (Actual); Study Completion 2017-06-18 (Actual)

PRIMARY OUTCOMES:
cardiorespiratory evaluation | 1 day
  a maximal treadmill test is proposed (evaluation of : VO² max, maximal heart rate)
autonomic nervous system evaluation | 1 day and 3 nights
  an orthostatic test is proposed in order to verify the ANS adaptation. A nocturnal recording is made during three nights in order to verify the possible link between the rest autonomic adaptations and a possible dysautonomia observed with the orthostatic test.
sleep evaluation | 7 nights
  Sleep characteristics are obtained by an actimetry during 7 nights in order to observe sleep disorders.
  Sleep Questionnaires are also completed.

SECONDARY OUTCOMES:
physical activity | 7 days
  physical activity characteristics (sedentary, moderate or vigorous activities, energy expenditure) are obtained by an actimetry during 7 days.
  Questionnaires of physical activity are also completed
Motor capacities | 1 day
  motor capacities are evaluated by several specific tests : PANESS, M-ABS and Eurofit.
Behavioural characteristics | 1 hour
  Behavioural characteristics are evaluated by the Vineland scale
biological parameters | 1 day
  during the maximal treadmill test, salivary samples are made (cortisol, alpha amylase), before and after tthe test

CONTACTS AND LOCATIONS:
Overall Officials: Véronique BRICOUT, PhD, Principal Investigator — CHU Grenoble France; Michel GUINOT, Dr, Principal Investigator — CHU Grenoble France
Locations (1):
- CHU Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No